CLINICAL TRIAL: NCT05247203
Title: A Phase I, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Telitacicept in Chinese Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Telitacicept Study in Chinese Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18C020
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Telitacicept; Pharmacokinetics; Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases | interventions — telitacicept; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Telitacicept Arm 1 (Experimental): Telitacicept 80mg, once a week for 24 weeks plus standard therapy
  Interventions: Biological: Telitacicept; Drug: standard therapy
- Telitacicept Arm 2 (Experimental): Telitacicept 160mg, once a week for 24 weeks plus standard therapy
  Interventions: Biological: Telitacicept; Drug: standard therapy
- Telitacicept Arm 3 (Experimental): Telitacicept 160mg, once a week for 12 weeks followed by once every two weeks for another 12 weeks plus standard therapy
  Interventions: Biological: Telitacicept; Drug: standard therapy
- Telitacicept Arm 4 (Experimental): Telitacicept 240mg, once a week for 24 weeks plus standard therapy
  Interventions: Biological: Telitacicept; Drug: standard therapy
- Telitacicept Arm 5 (Experimental): Telitacicept 240mg, once every two weeks for 24 weeks plus standard therapy
  Interventions: Biological: Telitacicept; Drug: standard therapy

INTERVENTIONS:
Biological: Telitacicept — subcutaneous injection
  Other Names: RC18
Drug: standard therapy — A standard regimen consists of the following medication(s) (alone or in combination)：corticosteroids, anti-malarials, non-steroidal anti-inflammatory drugs (NSAIDs), other immunosuppressive or immunomodulatory agents including azathioprine, mycophenolate mofetil, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine.

SUMMARY:
This is a multi-center, open-label, phase I study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetics, safety and efficacy of Telitacicept in Chinese patients with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who give consent to this study participation and sign informed consent form;
2. Males and females, between the ages of 18 and 65 years old, inclusive, at the screening visit;
3. Diagnosis of SLE as defined by the American College of Rheumatology (ACR) 1997 criteria, with 4 or more of the 11 ACR criteria present;
4. SELENA-SLEDAI score ≥8 points with a clinical SELENA-SLEDAI score ≥6 points if low complement levels and/or anti-ds-DNA antibodies are present at the screening visit;
5. Subjects with unequivocally positive test for anti-nuclear antibody (ANA) and/or anti-ds-DNA serum antibody;
6. Be on a SLE standard treatment regimen (and remain stable) for a period of at least 30 days prior to Day 0. The standard regimen consists of the following medication(s) (alone or in combination)：corticosteroids, anti-malarials, non-steroidal anti-inflammatory drugs (NSAIDs), other immunosuppressive or immunomodulatory agents including azathioprine, mycophenolate mofetil, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine.

Exclusion Criteria:

1. Subjects with severe lupus kidney disease (defined by proteinuria >6g/24h or serum creatinine >2.5mg/dL or serum creatinine >221μmol/L) or active nephritis requiring prohibited medications, or subjects requiring hemodialysis or prednisone (or its equivalent)≥100mg/d for a period of ≥14 days within 8 weeks of Day 0;
2. Central nervous system (CNS) disease associated with lupus or not [including seizures, psychosis, organic brain syndrome, cerebrovascular accident (CVA), encephalitis, CNS angiitis] within 8 weeks prior to the screening visit;
3. Laboratory abnormalities including, but not limited to the following:

   1. ALT/AST≥2×upper limit of normal (ULN);
   2. endogenous creatinine clearance rate<30 mL/min;
   3. white blood cell count<2.5×10^9/L;
   4. hemoglobin<85 g/L;
   5. platelet count<50×10^9/L;
4. Active hepatitis or a history of severe liver disease at the screening visit. Positive test for Hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibodies (HCVAb). If anti-HBcAb result is positive while HBsAg result is negative, hepatitis B virus (HBV)-(DNA) test will be performed. If HBV-DNA result is negative, the patient is eligible;
5. Subjects with immunodeficiency, uncontrolled severe infection or active/recurrent gastrointestinal ulcers;
6. Pregnant or lactating female subjects or sexually active subjects who refuse to practice the protocol-specified contraception throughout the study;
7. History of allergy to humanized biological products;
8. Subjects who received live vaccine within 28 days of Day 0;
9. Participation in any other investigational study drug trial in the past 28 days or 5 half-lives, whichever was longer, prior to Day 0. Subjects who participated in a clinical trial on B-cell-targeted drug, or tumor necrosis factor inhibitor, or interleukin receptor blocker within 12 months prior to Day 0 would be excluded;
10. Subjects who received other B-cell targeted drugs, such as Belimumab, rituximab or Epratuzumab within 12 months prior to Day 0;
11. Subjects who received tumor necrosis factor inhibitors, interleukin receptor blockers within 12 months prior to Day 0;
12. Subjects who received intravenous immune globulin (IVIG), or high dose prednisone or its equivalents (≥100mg/d) for a period of ≥ 14 days, or plasma exchange within 28 days prior to Day 0;
13. Subjects who received IL-2, Thalidomide, Tripterygium wilfordii or Chinese medicinal preparations containing Tripterygium wilfordii within 28 days prior to Day 0;
14. Subjects with active infections (herpes zoster, HIV infection, active tuberculosis, etc.) at the screening visit;
15. Subjects with depression or suicidal thoughts;
16. Any condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol..

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of Telitacicept | up to 42 days following the last dose of Telitacicept
  Cmax is defined as peak plasma concentration of Telitacicept
Time to reach Cmax (tmax) of Telitacicept | up to 42 days following the last dose of Telitacicept
  tmax is defined as time to reach Cmax of Telitacicept
Observed plasma concentration of Telitacicept just prior to the beginning of a dosing interval (Ctrough) | up to 42 days following the last dose of Telitacicept
  Ctrough is defined as observed plasma concentration of Telitacicept just prior to the beginning of a dosing interval
Average concentration (Cav) of Telitacicept | up to 42 days following the last dose of Telitacicept
  Average concentration of Telitacicept
Area under the curve from time zero to last quantifiable concentration (AUC 0-t) of Telitacicept | up to 42 days following the last dose of Telitacicept
  AUC 0-t is defined as area under the curve from time zero to last quantifiable concentration of Telitacicept
Area under the curve from time zero to tau (AUC 0-tau) of Telitacicept | up to 42 days following the last dose of Telitacicept
  AUC 0-tau is defined as area under the curve from time zero to tau of Telitacicept
Terminal elimination rate constant (λz) of Telitacicept | up to 42 days following the last dose of Telitacicept
  λz is defined as terminal elimination rate constant
Terminal elimination half-life (t1/2z) of Telitacicept | up to 42 days following the last dose of Telitacicept
  t1/2z is defined as terminal elimination half-life of Telitacicept
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) of Telitacicept | up to 42 days following the last dose of Telitacicept
  Vz/F is defined as apparent volume of distribution during the terminal phase after extravascular administration of Telitacicept
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of Telitacicept | up to 42 days following the last dose of Telitacicept
  CL/F is defined as apparent total body clearance of drug from plasma after extravascular administration of Telitacicept

SECONDARY OUTCOMES:
Percentage of participants achieving a SLE Responder Index (SRI) | Week 4, 8, 12, 16, 20, and 24
  Percentage of subjects with a ≥ 4 point reduction from baseline in SELENA-SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
Percentage of participants achieving a SELENA-SLEDAI improvement of ≥4 points | Week 4, 8, 12, 16, 20, and 24
  SELENA-SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105.
Change From Baseline to W24 in patient global assessment (PGA) | Week 4, 8, 12, 16, 20, and 24
  PGA is a visual analog scale scored from 0 to 3 (1=mild, 2=moderate, 3=severe).
Change From Baseline to W24 in IgG | Week 4, 8, 12, 16, 20, and 24
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline to W24 in IgA | Week 4, 8, 12, 16, 20, and 24
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline to W24 in IgM | Week 4, 8, 12, 16, 20, and 24
  Immunoglobulins (IgG, IgA and IgM) are proteins produced by plasma cells.
Change From Baseline to W24 in C3 | Week 4, 8, 12, 16, 20, and 24
  Complement (C3/C4) are proteins that are part of the immune system.
Change From Baseline to W24 in C4 | Week 4, 8, 12, 16, 20, and 24
  Complement (C3/C4) are proteins that are part of the immune system.
Number of Participants Experiencing Adverse Events (AEs) | up to 28 days following the last dose of Telitacicept
  Adverse event means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided